CLINICAL TRIAL: NCT02711839
Title: Office of Human Research, Taipei Medical University
Brief Title: Evaluation of White Sweet Potato Tube Feeding Formula on Type 2 Diabetic Residents in Long-term Care Institutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201505027
Record Dates: First submitted 2015-11-17; First posted 2016-03-17 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Commercial diabetic formula
  Interventions: Dietary Supplement: Commercial diabetic formula
- Treatment Group (Experimental): White sweet potato formula
  Interventions: Dietary Supplement: White sweet potato formula

INTERVENTIONS:
Dietary Supplement: Commercial diabetic formula — The formula were supplied 1500~1800 kcal daily depend on the patient's individual situation
  Other Names: diabetic formula
  Arms: Control Group
Dietary Supplement: White sweet potato formula — The formula were supplied 1500~1800 kcal daily depend on the patient's individual situation
  Other Names: White sweet potato
  Arms: Treatment Group

SUMMARY:
In order to response the increasing of aging population cause losing ability that need long-care needs, the project entitled "10-year long-term care program" from Executive Yuan in 2007 is carried out to assist economically disadvantaged and disabled elderly to acquire daily nutrition. Therefore, the long-term care resident's nutritional status got more attention than before. Out of control in blood glucose will not only increase bed sores and urinary tract infection in tube feeding residents but also rise medical expenditures. The nutritional status of long-term care institutions, anyang homes and nursing home are generally bad in nutrition management due to high cost of nutritional supplements from foreign imports that cause the burden of families. In this study, we will recruit diabetic subjects that divide into white sweet potato group (experimental group) and commercial formula group (control group) by using randomized, parallel and open clinical study through tube feeding in sixty days.

DETAILED DESCRIPTION:
All subjects will be evaluated the blood sugar and clinical nutrition assessment such as postural measurement, urine test and blood biomarker examination.

ELIGIBILITY:
Inclusion Criteria:

* Long-term stability nasogastric or gastrostomy-fed person.
* The physician diagnosed as diabetic and regular use of hypoglycemic drugs.

Exclusion Criteria:

* Psychosis or depression.
* Hba1c> 8.5%.
* High taking nutritional supplements or steroids drugs.
* Have undergone abdominal surgery caused by intestinal sticky.
* Suffering from cancer, ulcers, respiratory infections and other diseases.
* Currently receiving central venous nutrition therapy or intravenous nutrition therapy.
* Liver dysfunction (ALT ≧ 100 U / L), renal insufficiency (creatinine ≧ 3mg / dl), heart failure (NYFc II above), moderate anemia (hemoglobin <9 g / dl).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Han Lin, MS, Principal Investigator — Office of Human Research, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ooi CP, Loke SC. Sweet potato for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2013 Sep 3;2013(9):CD009128. doi: 10.1002/14651858.CD009128.pub3. PMID 24000051
- [Derived] Chen CM, Shih CK, Su YJ, Cheang KU, Lo SF, Li SC. Evaluation of white sweet potato tube-feeding formula in elderly diabetic patients: a randomized controlled trial. Nutr Metab (Lond). 2019 Oct 16;16:70. doi: 10.1186/s12986-019-0398-8. eCollection 2019. PMID 31636690

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 20 | 34
Completed | 16 | 24
Not Completed | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 16 | 24 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (5.7) | 68.9 (8.8) | 71.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: HbA1c After Intervention
Description: HbA1c value after 60 days intervention in both groups
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 24
percentage | 6.8 (1.1) | 6.4 (1.1)

2. Secondary Outcome: Albumin After Intervention
Description: Albumin value after 60 days intervention in both groups
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 24
g/dL | 3.4 (0.1) | 3.6 (0.3)

3. Secondary Outcome: Glucose After Intervention
Description: Glucose value after 60 days intervention in both groups
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 24
mg/dL | 126.7 (38.9) | 131.0 (45.4)

4. Secondary Outcome: Total Cholesterol After Intervention
Description: Total cholesterol value after 60 days intervention in both groups
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 24
mg/dL | 180.0 (53.6) | 150.1 (25.7)

5. Secondary Outcome: Triglyceride After Intervention
Description: Triglyceride value after 60 days intervention in both groups
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 16 | 24
mg/dL | 214.3 (112.2) | 145.4 (59.3)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the participants during intervention and assessed after 6 months.
Description: No adverse event was happened in participants.
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/24
Other Adverse Events (participants affected / at risk) | 0/16 | 0/24

LIMITATIONS AND CAVEATS:
Small experimental sample size and trial duration that may cause impose an obstacle in the detection of significant changes of the study measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No